CLINICAL TRIAL: NCT06211881
Title: Chidamide Combined With Gemcitabine, Vinorelbine, and Mitoxantrone Hydrochloride Liposome (Chi-GVM) Regimen for the Treatment of Relapsed/Refractory (R/R) Peripheral T-cell Lymphoma (PTCL) :A Multicenter, Open-label, Single-arm Study
Brief Title: Chi-GVM Regimen for the Treatment of R/R PTCL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-519
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Relapsed/Refractory Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chi-GVM (Experimental): Chi-GVM regimen (every 21 days is a treatment cycle):
  Chidamide 20 mg orally;gemcitabine 1g/m2, twice a week, intravenous infusion on day 1, vinorelbine 20 mg/m2, infusion on day 1; Mitoxantrone Hydrochloride Liposome12 mg/m2, intravenous infusion on day 1; Chidamide maintenance therapy: 20 mg orally twice a week/28 days/cycle.
  Interventions: Drug: Chi-GVM

INTERVENTIONS:
Drug: Chi-GVM — Chi-GVM regimen (every 21 days is a treatment cycle):
  Chidamide 20 mg orally;gemcitabine 1g/m2, twice a week, intravenous infusion on day 1, vinorelbine 20 mg/m2, infusion on day 1; Mitoxantrone Hydrochloride Liposome12 mg/m2, intravenous infusion on day 1; Chidamide maintenance therapy: 20 mg orally twice a week/28 days/cycle.
  Other Names: Chidamide Combined With Gemcitabine, Vinorelbine, and Mitoxantrone Hydrochloride Liposome

SUMMARY:
Peripheral T-cell lymphoma (PTCL) is a heterogeneous group of lymphoproliferative diseases caused by mature T cells, accounting for approximately 10% of non-Hodgkin lymphomas (NHL). PTCLs have a worse prognosis than aggressive B-cell lymphomas; they are less responsive to standard anthracycline-based chemotherapy regimens and responses are less durable. In an analysis of 341 patients with newly diagnosed PTCL who received anthracycline chemotherapy, 3-year PFS and OS rates were 32% and 52%, respectively, significantly inferior to matched patients with diffuse large B-cell lymphoma (DLBCL).And patients who received consolidative hematopoietic cell transplantation (HCT) had no significant benefit. The prognosis of relapsed/refractory (R/R) patients is even worse. Among the 420 evaluable R/R PTCL patients in the COMPLETE registration study, the median OS of R/R patients were 29 months and 12 months respectively . There is still no effective second-line regimen that can improve patient survival, so treatment options urgently need to be optimized.We designed a randomized, prospective, multi-center phase II clinical trial to explore the efficacy of chidamide combined with gemcitabine, vinorelbine and Mitoxantrone Hydrochloride Liposome (Chi-GVM) in the treatment of patients with R/R PTCL. We expected to further improve ORR, PFS and OS.

DETAILED DESCRIPTION:
Peripheral T-cell lymphoma (PTCL) is a heterogeneous group of lymphoproliferative diseases caused by mature T cells, accounting for approximately 10% of non-Hodgkin lymphomas (NHL). Peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS) is the most common subtype, accounting for approximately 26%. This was followed by angioimmunoblastic T-cell lymphoma (AITL; 19%), anaplastic large cell lymphoma (ALCL, ALK)-positive (7%), ALK-negative (6%), and enteropathy-associated T-cell lymphoma ( EATL) .

PTCLs have a worse prognosis than aggressive B-cell lymphomas; they are less responsive to standard anthracycline-based chemotherapy regimens and responses are less durable. In an analysis of 341 patients with newly diagnosed PTCL who received anthracycline chemotherapy, 3-year PFS and OS rates were 32% and 52%, respectively, significantly inferior to matched patients with diffuse large B-cell lymphoma (DLBCL).And patients who received consolidative hematopoietic cell transplantation (HCT) had no significant benefit. The prognosis of relapsed/refractory (R/R) patients is even worse. Among the 420 evaluable R/R PTCL patients in the COMPLETE registration study, the median OS of R/R patients were 29 months and 12 months respectively . There is still no effective second-line regimen that can improve patient survival, so treatment options urgently need to be optimized.

Histone deacetylase (HDAC) inhibitors such as belinostat, romidepsin, etc. have been confirmed to show good efficacy in R/R AITL;Chinise original drug Chidamide is mainly targeted at Class I HDAC inhibitors (HDACi) of HDAC subtypes 1, 2, and 3 and class IIb subtype 10 have the regulatory effect on abnormal epigenetic functions of tumors. It triggers chromatin remodeling by inhibiting related HDAC isoforms to increase the acetylation level of chromatin histones, resulting in changes in gene expression (ie, epigenetic changes) targeting multiple signaling pathways, thereby inhibiting tumor cells cycle, induce apoptosis of tumor cells, and at the same time have overall regulatory activity on cellular immunity, inducing and enhancing the tumor killing effect mediated by natural killer cells (NK) and antigen-specific cytotoxic T cells (CTL). Chidamide also induces tumor stem cell differentiation and reverses the epithelial-mesenchymal phenotypic transition (EMT) of tumor cells through epigenetic regulation mechanisms, thereby restoring the sensitivity of drug-resistant tumor cells to drugs and inhibiting tumor metastasis. play a potential role in recurrence and other aspects. The above unique mechanism of action characteristics lay the foundation for the combined application of chidamide and other chemotherapy drugs in tumor treatment. Its phase II clinical study explored the effectiveness and safety of chidamide monotherapy in patients with R/R PTCL. The objective response rate (ORR) assessed by the investigators was 29.1%, and the median duration of response (DOR) was 9.9 months, and is well tolerated.Chidamide has been included in the medical insurance indications for patients with relapsed or refractory PTCL who have received at least one systemic chemotherapy in the past. However, single drug is still not effective in patients with nTFHL and needs to be combined with other drugs.

Gemcitabine, dexamethasone, and cisplatin (GDP) combined with autologous hematopoietic stem cell transplantation (ASCT) can effectively treat patients with R/R PTCL, with an ORR of 72% to 80% and a CR of 47% to 48%. Among patients who subsequently underwent ASCT, 2-year post-transplant OS was 53%. A retrospective analysis showed that the gemcitabine, vinorelbine, and doxorubicin (GND) regimen was effective and well tolerated in patients with R/RT cell lymphoma (n=49; 28 patients with PTCL-NOS), with ORR was 65%, the median OS was 36 months, and the 5-year estimated OS rate was 32%.

ELIGIBILITY:
Inclusion Criteria:

* 1. R/R PTCL confirmed by pathological tissue [including peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), and ALK+ anaplastic large cell lymphoma (ALCL) , ALK-ALCL, monotypic epithelial intestinal T-cell lymphoma (MEITL), etc.], the diagnostic criteria refer to the 2022 WHO diagnostic criteria; 2. Have had at least one previous systemic treatment [including chemotherapy, autologous hematopoietic stem cell transplantation (ASCT) ), etc.] Patients who have no remission or relapse after remission; 3. Sign written informed consent and be able to comply with the visits and related procedures specified in the protocol; 4. Whole-body PET/CT performed 28 days before study enrollment must be At least 1 evaluable or measurable lesion that meets the Lugano2014 criteria: lymph node lesions, measurable lymph nodes must have a long diameter >1.5 cm; non-lymph node lesions, measurable extranodal lesions must have a long diameter >1.0 cm; 5. ECOG PS score: 0~2; 6. Have adequate organ and bone marrow function, defined as follows: neutrophil count ≥1.5×109/L, platelet count ≥75×109/L, hemoglobin ≥80 g/L (neutrophil count in patients with bone marrow involvement) The granulocyte count can be relaxed to ≥1.0×109/L, the platelet count can be relaxed to ≥50×109/L, and the hemoglobin can be relaxed to ≥75 g/L); 7. Liver and renal function: Serum creatinine (Cr) ≤1.5 times the upper limit of normal values; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal values (≤5 times the upper limit of normal values for patients with liver invasion); total bilirubin (TBIL) ) ≤ 1.5 times the upper limit of normal value (for patients with liver invasion ≤ 3 times the upper limit of normal value); 8. Expected survival time more than 3 months; 9. Age 18~75 years old.

Exclusion Criteria:

* 1. The subject's previous anti-tumor treatment history meets one of the following conditions:

  1. Those who have received mitoxantrone or Mitoxantrone Hydrochloride Liposome in the past;
  2. Previously received treatment with doxorubicin or other anthracyclines, with a total cumulative dose of doxorubicin >360 mg/m2 (converted from other anthracyclines, 1 mg of doxorubicin is equivalent to 2 mg of epirubicin );
  3. Patients who have received ASCT within 100 days of first medication, or have received allogeneic hematopoietic stem cell transplantation (Allo-SCT);
  4. Within 4 weeks before using this study drug for the first time, you have received anti-tumor treatment (including chemotherapy, targeted therapy, hormone therapy, taking traditional Chinese medicine with anti-tumor activity, etc.) or participated in other clinical trials and received clinical trial drugs.

  2. Have a hypersensitivity reaction to any study drug or its ingredients; 3. Uncontrollable systemic diseases (such as advanced infection, uncontrollable hypertension, diabetes, etc.); 4. Heart function and disease meet one of the following conditions:
  1. Long QTc syndrome or QTc interval >480 ms;
  2. Complete left bundle branch block, II or III degree atrioventricular block;
  3. Severe, uncontrolled arrhythmia requiring drug treatment;
  4. New York Heart Association classification ≥ III;
  5. The cardiac left ventricular ejection fraction (LVEF) is less than 50%;
  6. Have a history of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, clinically severe pericardial disease, or acute ischemic or active disease within 6 months before recruitment Electrocardiographic evidence of sexual conduction system abnormalities.

  5. Active infection of hepatitis B and hepatitis C (hepatitis B virus surface antigen is positive and hepatitis B virus DNA exceeds 1×103 copies/mL; hepatitis C virus RNA exceeds 1×103 copies/mL); 6. Human immunodeficiency virus (HIV) infection (HIV antibody positive); 7. Have suffered from other malignant tumors in the past or at the same time (except for non-melanoma basal cell carcinoma of the skin, breast/cervical carcinoma in situ and other malignant tumors that have been effectively controlled without treatment in the past 5 years); 8. Suffer from primary or secondary central nervous system (CNS) lymphoma or have a history of CNS lymphoma at the time of recruitment; 9. Pregnant, lactating women and patients of childbearing age who are unwilling to take contraceptive measures; 10. People with mental disorders/people unable to obtain informed consent; 11.Those who are judged by the researcher to be unsuitable to participate in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  overall response rate

SECONDARY OUTCOMES:
DoR | 2 years
  Duration of Response
2-years OS | 2 years
  2-year overall survival
2-years PFS | 2 years
  2-year progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: wei Xu, Doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu, China